CLINICAL TRIAL: NCT03687021
Title: Clinical Study on the Impact of Route of Administration of Progesterone and Endometriosis on Endometrial Receptivity
Brief Title: Clinical Study on Endometrial Receptivity
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: yuqi03029
Record Dates: First submitted 2018-08-13; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-08

CONDITIONS: Endometrial Receptivity;RNA; Progesterone
Keywords: endometrial receptivity; RNA; progesterone
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- endometriosis (No Intervention): tissue biopsy from patients (n=10) with endometriosis
- without endometriosis (No Intervention): tissue biopsy from patients (n=10) without endometriosis
- Intramuscular progesterone (Experimental): Intramuscular progestin(20mg)
  Interventions: Drug: Progesterone
- vaginal progesterone (Experimental): vaginal progestin (90mg)
  Interventions: Drug: Progesterone
- oral progesterone (Experimental): oral progestin(40mg)
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — Different routes of administration of progesterone; Whether there is endometriosis
  Arms: Intramuscular progesterone; oral progesterone; vaginal progesterone

SUMMARY:
to explore the differential expression of miRNA in the implantation window of patients with endometriosis and the time of progesterone and route of administration on planting window

ELIGIBILITY:
Inclusion Criteria:

1. The endometriosis group treatment group: Previous laparoscopy or laparotomy confirmed endometriosis;Regular menstruation, no rule vaginal bleeding;Ovarian reserve function is normal.

   control group: Laparoscopic bilateral salpingectomy was performed due to ectopic pregnancy, benign ovarian changes and other reasons, with the exception of endometriosis during the operation.Regular menstruation, no rule vaginal bleeding;Ovarian reserve function is normal
2. progesterone group Women with hypothalamic amenorrhea or premature ovarian failure;Ages 18-40

Exclusion Criteria:

Patients with medical complications

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-10-10 (Estimated); Primary Completion 2018-10-10 (Estimated); Study Completion 2018-11-10 (Estimated)

PRIMARY OUTCOMES:
endometrial receptivity measured by pathology | 3 months
  35 samples will be measured.

SECONDARY OUTCOMES:
endometrial receptivity measured by immunohisochemistry | 3 months
  35 samples will be measured
endometrial receptivity measured by Ribose Nucleic Acid （RNA） | 3 months
  35 samples will be measured
endometrial receptivity measured by scanning electron microscope | 3 months
  35 samples will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Peking Union Medical College and Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No